CLINICAL TRIAL: NCT05088603
Title: The Effect of Clear Masks on Patient Satisfaction With Physician Communication During Awake Brain Surgery
Brief Title: Effect of Clear Masks on Patient Satisfaction With Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00077199
Record Dates: First submitted 2021-10-13; First posted 2021-10-22 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2023-09

CONDITIONS: Communication; Patient Satisfaction
Keywords: clear mask; neurological condition; deep brain stimulation; brain surgery; neurology
MeSH Terms: conditions — Communication; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: The neurologist will wear the mask type assigned by randomization for the duration of involvement in the surgery. At the conclusion of the neurologist's interaction with the participant, the participant will be asked a series of questions to evaluate the communication experience. This step will be performed by another member of the study team (not the participating neurologist) who will read from the questionnaire and record the participant's responses. During questioning, the neurologist will step out of the operating room to reduce potential bias from the participants answering subjective questions in front of the neurologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Clear Mask (Experimental): Subjects randomized to this group will have a neurologist who wears a clear mask during their procedure and during their interaction with the subject.
  Interventions: Device: Clear Mask
- Standard Mask (No Intervention): Subjects randomized to this group will have a neurologist who wears a standard mask during their procedure and during their interaction with the subject.

INTERVENTIONS:
Device: Clear Mask — The clear mask has a 4.75 x 1.35 inch clear window that allows for clear visibility of the mouth.
  Arms: Clear Mask

SUMMARY:
The purpose of this research study is to evaluate participants' experience and satisfaction during the awake deep brain stimulation (DBS) procedure. Normally, the neurologist will ask the participant questions and also ask the participant to perform tasks during surgery. During this time, the neurologist will be talking to the participant and the participant will be responding by answering questions or participating with the tasks.

For some study participants, there will be one small change made to the typical way the neurologist conducts this evaluation. The study staff will then ask the study participants about their experience with the neurologist's evaluation. The subject will not be told what part of the evaluation is changed for the study, until after they have responded to the questionnaire.

DETAILED DESCRIPTION:
All participants scheduled for a DBS phase I surgery will be contacted via telephone in the days prior to their scheduled surgery to discuss the possibility of study participation. This will be done to give the participant time to consider study participation in order to avoid delays the morning of surgery. The morning of surgery the participant will be approached in pre-operative holding room to discuss participation in the study and if amenable sign consent for participation. This discussion will inform the participant that minor changes are being made in an attempt to improve the participant experience, but limited information will be shared to reduce potential bias that might result from the participant knowing what is being studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients electing to undergo deep brain stimulator placement
* Patient in whom general anesthesia is not planned for stimulator target localization

Exclusion Criteria:

* Patients who do not give consent
* Patients who do not undergo DBS placement
* Patients who are blind or have a severe visual impairment
* Non-English speaking patients (i.e., patients for whom an interpreter would be needed to conduct the intra-operative assessment)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Hsu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clear Mask | Standard Mask
Started | 37 | 35
Completed | 31 | 34
Not Completed | 6 | 1
Not completed — Protocol Violation | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clear Mask | Standard Mask | Total
Number analyzed (Participants) | 31 | 34 | 65
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69.0 [55.0 to 72.0] | 68.5 [63.0 to 75.0] | 69.0 [60.0 to 73.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 19 | 28 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White, non-Hispanic | 31 | 33 | 64
  Race/Ethnicity: Unknown/Not Reported | 0 | 1 | 1
Indication for DBS [Count of Participants; unit: Participants]
  Dystonia | 3 | 0 | 3
  Essential Tremor | 9 | 12 | 21
  Parkinson's Disease | 19 | 22 | 41
HHIE -S Overall Score [Median (Inter-Quartile Range); unit: units on a scale] — Hearing Handicap Inventory - Screening Version. Total score was sum of points across 10 questions. Responses were "No" (0 points), "Sometimes" (2 points) or "Yes" (4 points). Interpretation of Total Score: 0-8 = no handicap; 10-24 = mild to moderate handicap; 26-40 = severe handicap
  units on a scale | 0 [0 to 10] | 7 [0 to 14.5] | 4 [0 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Positive Response Score of 4 to Question 1 on the Clinician & Group Survey-Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS) Questionnaire
Description: Questionnaire measures the subject's satisfaction and experience with his or her physician and/or physician practice. Question #1 of the CG-CAHPS is "Did this provider explain things in a way that was easy to understand?" with 1 meaning "not at all" and 4 meaning "completely". Responses 1-3 were considered negative and response 4 considered positive. Outcome is count of positive responses.
Time Frame: Day 1 Post Surgery
Population: All randomized subjects who were not excluded due to a protocol deviation.
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Mask | Standard Mask
Number analyzed (Participants) | 31 | 34
Participants | 29 | 29
Statistical Analysis 1: Comparison: Clear Mask vs Standard Mask; Test type: Superiority; p = 0.106, Fisher Exact

2. Secondary Outcome: Number of Participants With a Positive Response Score of 4 to Question 2 on the Clinician & Group Survey-Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS) Questionnaire
Description: Questionnaire measures the subject's satisfaction and experience with his or her physician and/or physician practice. Question 2 "Did this provider listen carefully to you?" with 1 meaning "not at all" and 4 meaning "completely". Responses 1-3 were considered negative and response 4 considered positive. Outcome is count of positive responses.
Time Frame: Day 1 Post Surgery
Population: All randomized subjects who were not excluded due to a protocol deviation
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Mask | Standard Mask
Number analyzed (Participants) | 31 | 34
Participants | 31 | 33
Statistical Analysis 1: Comparison: Clear Mask vs Standard Mask; Test type: Superiority; p = 0.99, Fisher Exact

3. Secondary Outcome: Number of Participants With a Positive Response Score of 4 to Question 3 on the Clinician & Group Survey-Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS) Questionnaire
Description: Questionnaire measures the subject's satisfaction and experience with his or her physician and/or physician practice. Question 3 "Did this provider seem to know the important information about your medical history?" with 1 meaning "not at all" and 4 meaning "completely". Responses 1-3 were considered negative and response 4 considered positive. Outcome is count of positive responses.
Time Frame: Day 1 Post Surgery
Population: Missing one participant response to this question
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Mask | Standard Mask
Number analyzed (Participants) | 30 | 34
Participants | 28 | 32
Statistical Analysis 1: Comparison: Clear Mask; Test type: Superiority; p = 0.99, Fisher Exact

4. Secondary Outcome: Number of Participants With a Positive Response Score of 4 to Question 4 on the Clinician & Group Survey-Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS) Questionnaire
Description: Questionnaire measures the subject's satisfaction and experience with his or her physician and/or physician practice. Question 4 "Did this provider show respect for what you had to say?" with 1 meaning "not at all" and 4 meaning "completely". Responses 1-3 were considered negative and response 4 considered positive. Outcome is count of positive responses.
Time Frame: Day 1 Post Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Mask | Standard Mask
Number analyzed (Participants) | 31 | 34
Participants | 31 | 34

5. Secondary Outcome: Number of Participants With a Positive Response Score of 4 to Question 5 on the Clinician & Group Survey-Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS) Questionnaire
Description: Questionnaire measures the subject's satisfaction and experience with his or her physician and/or physician practice. Question 5 "Did this provider spend enough time with you?" with 1 meaning "not at all" and 4 meaning "completely". Responses 1-3 were considered negative and response 4 considered positive. Outcome is count of positive responses.
Time Frame: Day 1 Post Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Mask | Standard Mask
Number analyzed (Participants) | 31 | 34
Participants | 31 | 32
Statistical Analysis 1: Comparison: Clear Mask vs Standard Mask; Test type: Superiority; p = 0.529, Fisher Exact

6. Secondary Outcome: Number of Participants With a Positive Response Score of 4 to Question 6 on the Clinician & Group Survey-Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS) Questionnaire
Description: Questionnaire measures the subject's satisfaction and experience with his or her physician and/or physician practice. Question 6 "Did this provider demonstrate empathy?" with 1 meaning "not at all" and 4 meaning "completely". Responses 1-3 were considered negative and response 4 considered positive. Outcome is count of positive responses.
Time Frame: Day 1 Post Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Mask | Standard Mask
Number analyzed (Participants) | 31 | 34
Participants | 29 | 32
Statistical Analysis 1: Comparison: Clear Mask vs Standard Mask; Test type: Superiority; p = 0.99, Fisher Exact

7. Secondary Outcome: Number of Participants With a Positive Response Score of 4 to Question 7 on the Clinician & Group Survey-Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS) Questionnaire
Description: Questionnaire measures the subject's satisfaction and experience with his or her physician and/or physician practice. Question 7 "How comfortable do you feel trusting the provider's decisions?" with 1 meaning "not at all" and 4 meaning "completely". Responses 1-3 were considered negative and response 4 considered positive. Outcome is count of positive responses.
Time Frame: Day 1 Post Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Mask | Standard Mask
Number analyzed (Participants) | 31 | 34
Participants | 29 | 29
Statistical Analysis 1: Comparison: Clear Mask vs Standard Mask; Test type: Superiority; p = 0.502, Fisher Exact

8. Secondary Outcome: Number of Participants With a Positive Response Score of 4 to Question 8 on the Clinician & Group Survey-Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS) Questionnaire
Description: Questionnaire measures the subject's satisfaction and experience with his or her physician and/or physician practice. Question 8 "Did you understand what you were being asked to do?" with 1 meaning "not at all" and 4 meaning "completely". Responses 1-3 were considered negative and response 4 considered positive. Outcome is count of positive responses.
Time Frame: Day 1 Post Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Mask | Standard Mask
Number analyzed (Participants) | 30 | 34
Participants | 29 | 30
Statistical Analysis 1: Comparison: Clear Mask vs Standard Mask; Test type: Superiority; p = 0.431, Fisher Exact

9. Secondary Outcome: Number of Participants With a Positive Response Score of 4 to Question 9 on the Clinician & Group Survey-Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS) Questionnaire
Description: Questionnaire measures the subject's satisfaction and experience with his or her physician and/or physician practice. Question 9 "How satisfied are you with the procedure thus far overall?" with 1 meaning "not at all" and 4 meaning "completely". Responses 1-3 were considered negative and response 4 considered positive. Outcome is count of positive responses.
Time Frame: Day 1 Post Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Mask | Standard Mask
Number analyzed (Participants) | 31 | 34
Participants | 27 | 26
Statistical Analysis 1: Comparison: Clear Mask vs Standard Mask; Test type: Superiority; p = 0.434, Fisher Exact

10. Secondary Outcome: Number of Participants With a Positive Response Score of 4 to Question 10 on the Clinician & Group Survey-Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS) Questionnaire
Description: Participants were asked "What was your impression of the doctor's mask" with 1 meaning "Strongly Disliked" and 4 meaning "Strongly Liked". Responses 1-3 were considered negative and response 4 considered positive. Outcome is count of positive responses.
Time Frame: Day 1 Post Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Mask | Standard Mask
Number analyzed (Participants) | 26 | 30
Participants | 20 | 17
Statistical Analysis 1: Comparison: Clear Mask vs Standard Mask; Test type: Superiority; p = 0.159, Fisher Exact

11. Secondary Outcome: Number of Participants With a Positive Response to Question 11 on the Clinician & Group Survey-Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS) Questionnaire
Description: Participants were asked "What comments do you have about the doctor's mask." The free text responses were categorized as positive/negative/neutral. Outcome is count of positive responses.
Time Frame: Day 1 Post Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Mask | Standard Mask
Number analyzed (Participants) | 31 | 34
Participants | 9 | 2
Statistical Analysis 1: Comparison: Clear Mask vs Standard Mask; Test type: Superiority; p = 0.051, Fisher Exact

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Clear Mask | Standard Mask
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/34
Other Adverse Events (participants affected / at risk) | 0/31 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT05088603/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT05088603/ICF_000.pdf